CLINICAL TRIAL: NCT07058220
Title: Physical Therapist at 23 July Hospital Marg Egypt
Brief Title: Effect Cervical Proprioceptive Training Cervical Proprioception Neck Pain:
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma eldesoky, Senior physical therapist at sadr El-Marg hospital Cairo Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No:SREC.PT.SUE(5)325
Record Dates: First submitted 2025-05-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Cervical Joint Position Error; Cervical Pain
Keywords: neck pain; cervical proprioception; training; exercise; proprioceptive error
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive training group (Experimental)
  Interventions: Other: Advices
- Conventional group (Active Comparator)
  Interventions: Other: Cervical proprioceptive training

INTERVENTIONS:
Other: Cervical proprioceptive training — Study group will receive proprioceptive training through use of a laser pointer in a similar way to the testing. From sitting position, patients were asked to flex, extend and rotate their head and then return to the neutral position . This training was commenced with open eyes. Each direction was repeated 8 times for two sets, 30 seconds rest between sets. Progression of exercise was achieved by closing eyes, and altering the duration (trace shapes for 5 minutes and progress by increasing 2-3 minutes weekly as tolerated), repetitions (2-3 repetitions weekly), sets (1 set weekly) and the degree of difficulty of the task (different shapes and positions as standing and walking)
  Arms: Conventional group
Other: Advices — Patients of control group were allowed to stay active, avoid poor cervical ergonomics (poor sleeping habits, improper use of mobile/telephone),hot/cold packs, some range of motion exercises, and local medicines as prescribed by their general practitioner.
  Arms: Proprioceptive training group

SUMMARY:
Twenty-two male and female patients with neck pain participated in this study, aged from 25-40 years. They randomly distributed into 2 group: group (A, study) consisted of 11 patients received cervical proprioceptive training, while group (B, control) consisted of 11 patients received usual care. The treatment was performed 3 times per week for 1 month. The cervical proprioception (flexion, extension, right and left rotations) was assessed by Revel laser method as active joint angular reproduction [absolute error].

DETAILED DESCRIPTION:
Twenty-two male and female patients referred from orthopedist. Patients were selected in the study if they had non-specific neck pain, aged from 25-40 years. Patients were excluded if they had positive spurling test.

All patients were randomly distributed into two groups. Group (A) or study group consisted of 11 patients received cervical proprioceptive training, while group (B) or control group consisted of 11 patients received standard care. The treatment was performed 3 times per week for 1 month. The cervical proprioception [active joint angular reproduction, absolute error] assessed by revel laser method.

Laser pointer" was used for assessing cervical proprioception. It had good reliability (r=0.68) and validity (r=0.95). The patient sat with back supported and head free to move. The target paper was fixed on the wall about 90 cm from the seat and at a distance from the ground adjusted with the height of the patient. A "laser pointer" was strapped on the highest point of the head of the patient. The patient was instructed to move the head to the tested direction (flexion and extension, and right and left rotation), then fix the laser beam at the paper center for 10 seconds while opening the eyes. The reached point in each direction was marked. Then the distance between the paper center and the reached point was measured using a tape measurement

Treatment procedures:

Cervical proprioceptive training (CPT): patients of group A received CPT through use of a laser pointer in a similar way to the testing. From sitting position, patients were asked to flex, extend and rotate their head and then return to the neutral position . This training was commenced with open eyes. Each direction was repeated 8 times for two sets, 30 seconds rest between sets. Progression of exercise was achieved by closing eyes, and altering the duration (trace shapes for 5 minutes and progress by increasing 2-3 minutes weekly as tolerated), repetitions (2-3 repetitions weekly), sets (1 set weekly) and the degree of difficulty of the task (different shapes and positions as standing and walking) .

Standard care: Patients of control group were allowed to stay active, avoid poor cervical ergonomics (poor sleeping habits, improper use of mobile/telephone),hot/cold packs, some range of motion exercises, and local medicines as prescribed by their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* they had non-specific neck pain

Exclusion Criteria:

* they had positive spurling test.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cervical joint position error error | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo y, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No